CLINICAL TRIAL: NCT05879861
Title: Development and Validation of a Risk Prediction Model for Preoperative Frailty in Elderly Patients With Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Yongmei Zhang, Study Director, Zunyi Medical College
Other Study IDs: ZSKHZ Zi (2022) no. 337
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fried Scale and its related scales were used to analyze the status and risk factors of preoperative frailty in elderly patients with colorectal cancer. R software was used to construct a risk prediction model for preoperative frailty in elderly patients with colorectal cancer, and its validity and stability were verified in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. patients who met the diagnostic criteria of colorectal cancer in Chinese Guidelines for Diagnosis and Treatment of Colorectal Cancer 2020 Edition and underwent surgery;
2. patients aged ≥60 years old ;
3. patients who are clearly conscious, able to understand instructions, communicate normally, and complete the physical activity ability test without the assistance of others;
4. patients who gave informed consent and volunteered to participate in the study.

Exclusion Criteria:

1. patients with limb joint disease and lower limb pain;
2. patients with serious heart, liver, kidney diseases could not complete the test;
3. patients with visual impairment and hearing impairment;
4. patients with a history of mental illness or drug dependence;
5. taking antidepressants, levodopa/carbidopa, donepezil hydrochloride and other drugs ;
6. patients who received preoperative radiotherapy and chemotherapy;
7. Patients with hypothyroidism, Parkinson's disease, stroke and other diseases.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who met the diagnostic criteria of colorectal cancer in Chinese Guidelines for Diagnosis and Treatment of Colorectal Cancer 2020 Edition and underwent surgery.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Status of frailty | 1 day
  Status of frailty will be assessed by Fried Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Zhang, Study Director — Zunyi Medical College
Locations (1):
- Yongmei Zhang, Zunyi, Guizhou, China